CLINICAL TRIAL: NCT02915770
Title: Clinical Application of Cholangiojejunostomy in the Surgical Treatment of Cholelithiasis With Moderate Dilatation of Common Bile Duct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Dajiang li, associate professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014（18）
Record Dates: First submitted 2016-07-06; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Cholangiojejunostomy; Cholelithiasis
Keywords: Moderate dilatation of common bile duct
MeSH Terms: conditions — Cholelithiasis | interventions — Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- participants receive cholangiojejunostomy (Experimental): participants will receive hepatectomy、cholangiojejunostomy and T-tube Drainage
  Interventions: Procedure: cholangiojejunostomy; Procedure: hepatectomy; Device: T-tube
- participants receive no cholangiojejunostomy (Active Comparator): participants will receive hepatectomy and T-tube Drainage
  Interventions: Procedure: hepatectomy; Device: T-tube

INTERVENTIONS:
Procedure: cholangiojejunostomy — Half of participants will receive hepatectomy, cholangiojejunostomy and T-tube Drainage,while the other half will receive hepatectomy and T-tube Drainage
  Arms: participants receive cholangiojejunostomy
Procedure: hepatectomy
Device: T-tube — T-tube Drainage

SUMMARY:
This study evaluates the clinical application of cholangiojejunostomy in the surgical treatment of cholelithiasis with Moderate dilatation of common bile duct. Half of participants will receive hepatectomy, cholangiojejunostomy and T-tube Drainage, while the other half will receive hepatectomy and T-tube Drainage.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic bile duct stone disease, need surgery
* No residual stones in the operation
* Extrahepatic bile duct dilatation, 15-30 mm in diam.
* No relaxation or stenosis of the sphincter of Oddi

Exclusion Criteria:

* Patient involuntary
* Surgical treatment can not be performed because of various reasons.
* Intrahepatic and extrahepatic bile duct stones can not be taken away
* with other biliary tract diseases, such as bile duct cancer
* Oddi sphincter relaxation or stenosis
* loss to follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence of bile duct stones | 2-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatobiliary Surgery Institute, Southwest Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided